CLINICAL TRIAL: NCT02404103
Title: Flunisolide HFA in Children With Small Airway Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Meda Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Nemr Eid, Principal investigator, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14.1024
Record Dates: First submitted 2015-03-18; First posted 2015-03-31 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-11

CONDITIONS: Childhood Asthma
MeSH Terms: interventions — flunisolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flunisolide 160 mcg per day (Active Comparator): Patients will receive inhaled Flunisolide HFA 80 mcg twice per day for a total of 160 mcg per day over the 6 week study period
  Interventions: Drug: Flunisolide HFA
- Flunisolide 320 mcg per day (Active Comparator): Patients will receive inhaled Flunisolide HFA 160 mcg twice per day for a total of 320 mcg per day over the 6 week study period
  Interventions: Drug: Flunisolide HFA

INTERVENTIONS:
Drug: Flunisolide HFA

SUMMARY:
The purpose of this study is to see how two doses of Flunisolide HFA (an FDA approved inhaled medication to treat asthma) affect the small airways in children with asthma.

DETAILED DESCRIPTION:
This is a prospective, randomized, parallel, open label study. The primary aim is to compare the average change in spirometric values (Forced expiratory volume 1 (FEV1) and Forced Expiratory Flow 25-75% (FEF 25-75%) and Impulse Oscillometry System (IOS) values (Resistance at 5 Hz (R5), Resistance at 20 Hz (R20), Area of reactance (AX), Resonant frequency (Fres)) from baseline to week 6 from participants randomized flunisolide hydrofluoroalkane (HFA) 1 inhalation BID and to flunisolide HFA 2 inhalations BID. The change in scores from baseline to six week follow up will initially be compared using paired t-tests and Chi-squared tests for trend. Repeated measurements will be analyzed using generalized linear mixed-effects regression modeling (GLMM) techniques. For continuous outcomes (e.g. FEV1, FEF 25-75%, Fres, reactance at 5 Hz (X5), AX, R5-R20). The identity link function and normal distribution will be used. For count data (e.g., use of Beta-agonists, episodes of coughing, episodes of wheezing, etc.) the log link function and the Poisson distribution will be used. If we dichotomize outcomes (e.g., a Beta-agonist was used, coughing occurred, etc.) the logit link function and Bernoulli distribution will be used.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Informed consent by parent or legal guardian
* 6 years to 18 years of age at screening visit
* ability to comply with medication use, study visits and study procedures as judged by the site investigator
* FEF 25-75% <65% of predicted as a marker for small airway disease

Exclusion Criteria:

* Acute wheezing at screening visit or at Baseline visit
* Acute intercurrent respiratory infection, defined as an increase in cough, wheezing, or respiratory rate with onset in 1 week preceding screening visit or 3 weeks preceding baseline visit
* Oxygen saturation <95% at screening visit or at Baseline visit
* Clinically significant upper airway obstruction as determined by the Site Investigator (e.g. severe laryngomalacia, markedly enlarged tonsils, significant snoring, diagnosed obstructive sleep apnea.
* Severe gastroesophageal reflux, defined as persistent frequent emesis despite anti-reflux therapy
* Physical findings that would compromise the safety of the subject or the quality of the study data as determined by site investigator
* Inhaled Corticosteroids (ICS) use within 7 days of Baseline visit; systemic steroids within 30 days
* Cystic Fibrosis, Interstitial lung disease (ILD) history of severe Bronchopulmonary dysplasia (BPD) or other underling significant respiratory disease apart from asthma
* Potential subjects who are pregnant may not enroll in the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2015-03; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville Pediatric Pulmonology, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Flunisolide 160 mcg Per Day: Patients will receive inhaled Flunisolide HFA 80 mcg twice per day for a total of 160 mcg per day over the 6 week study period
  Flunisolide HFA
- Flunisolide 320 mcg Per Day: Patients will receive inhaled Flunisolide HFA 160 mcg twice per day for a total of 320 mcg per day over the 6 week study period
  Flunisolide HFA
Period: Overall Study
Arm/Group | Flunisolide 160 mcg Per Day | Flunisolide 320 mcg Per Day
Started | 14 | 12
Completed | 10 | 9
Not Completed | 4 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Population: Those subjects that completed the study protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Flunisolide 160 mcg Per Day | Flunisolide 320 mcg Per Day | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (3.8) | 11.1 (2.9) | 10.5 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Spirometry Forced Expiratory Volume 1 (FEV1) After Flunisolide
Description: the most used outcome in respiratory studies
Time Frame: Before and after treatment at baseline and six week followup
Population: Those subjects that completed the study protocol.
Measure: Mean (Standard Deviation); unit: % of predicted
Groups:
- Flunisolide 160 mcg Per Day Pretreatment - Baseline: Baseline value for Patients who received inhaled Flunisolide HFA 80 mcg twice per day for a total of 160 mcg per day over the 6 week study period
  Flunisolide HFA
- Flunisolide 320 mcg Per Day Pretreatment - Baseline: Baseline for patients who received inhaled Flunisolide HFA 160 mcg twice per day for a total of 320 mcg per day over the 6 week study period
  Flunisolide HFA
- Flunisolide 160 mcg Per Day Posttreatment - 6 Wks: After 6 weeks treatment value for Patients who received inhaled Flunisolide HFA 80 mcg twice per day for a total of 160 mcg per day over the 6 week study period
- Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks: After 6 week valeus for patients who received inhaled Flunisolide HFA 160 mcg twice per day for a total of 320 mcg per day over the 6 week study period
  Flunisolide HFA
Arm/Group | Flunisolide 160 mcg Per Day Pretreatment - Baseline | Flunisolide 320 mcg Per Day Pretreatment - Baseline | Flunisolide 160 mcg Per Day Posttreatment - 6 Wks | Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks
Number analyzed (Participants) | 10 | 9 | 10 | 9
% of predicted | 80.4 (10.8) | 78.7 (9.0) | 85.0 (10.3) | 77.0 (7.6)
Statistical Analysis 1: Comparison: Flunisolide 160 mcg Per Day Posttreatment - 6 Wks vs Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks; Test type: Equivalence — The primary goal of the current study is to determine the effects of Aerospan on lung function in children with small airway obstruction with two doses; p = .148, Mixed Models Analysis; generalized linear mixed-effects models (GLMM) using the identity link function and normal distribution were used
Statistical Analysis 2: Comparison: Flunisolide 160 mcg Per Day Pretreatment - Baseline vs Flunisolide 160 mcg Per Day Posttreatment - 6 Wks; Test type: Equivalence — A goal was to evaluate whether flunisolide HFA 320 mcg when compared to flunisolide 160 mcg lead to significantly better improvement in the same outcome measures over time; p = .740, Mixed Models Analysis
Statistical Analysis 3: Comparison: Flunisolide 320 mcg Per Day Pretreatment - Baseline vs Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks; Test type: Equivalence — generalized linear mixed-effects models (GLMM) using the identity link function and normal distribution were used; p = .921, Mixed Models Analysis

2. Primary Outcome: Impulse Oscillometry (IOS) Area of Reactance (AX) After Flunisolide Treatment
Description: A composite measure of small airway dysfunction. A reduction in IOS scores indicate an improvement.
Time Frame: Baseline and six week followup
Population: Those subjects that completed the study protocol.
Measure: Mean (Standard Deviation); unit: cmH2O/L
Groups:
- Flunisolide 160 mcg Per Day Pretreatment - Baseline: Before Patients received inhaled Flunisolide HFA 80 mcg twice per day for a total of 160 mcg per day over the 6 week study period
  Flunisolide HFA
- Flunisolide 320 mcg Per Day Pretreatment - Baseline: Before Patients received inhaled Flunisolide HFA 160 mcg twice per day for a total of 320 mcg per day over the 6 week study period
  Flunisolide HFA
- Flunisolide 160 mcg Per Day Posttreatment - 6 Wks: After 6 weeks treatment value forPatients who received inhaled Flunisolide HFA 80 mg twice per day.
- Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks: After 6 weeks treatment value for Patients who received inhaled Flunisolide HFA 160 mg twiece a day.
Arm/Group | Flunisolide 160 mcg Per Day Pretreatment - Baseline | Flunisolide 320 mcg Per Day Pretreatment - Baseline | Flunisolide 160 mcg Per Day Posttreatment - 6 Wks | Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks
Number analyzed (Participants) | 10 | 9 | 10 | 9
cmH2O/L | 17.4 (12.3) | 13.9 (16.6) | 18.5 (9.6) | 14.9 (13.5)
Statistical Analysis 1: Comparison: Flunisolide 160 mcg Per Day Pretreatment - Baseline vs Flunisolide 160 mcg Per Day Posttreatment - 6 Wks; Test type: Equivalence — The primary goal of the current study is to determine the effects of Aerospan on lung function in children with small airway obstruction; p = .872, Mixed Models Analysis; generalized linear mixed-effects models (GLMM) using the identity link function and normal distribution were used
Statistical Analysis 2: Comparison: Flunisolide 160 mcg Per Day Posttreatment - 6 Wks vs Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks; Test type: Equivalence — secondary goal was to evaluate whether flunisolide HFA 320 mcg when compared to flunisolide 160 mcg lead to significantly better improvement in the same outcome measures over time; p = 0.820, Mixed Models Analysis; generalized linear mixed-effects models (GLMM) using the identity link function and normal distribution were used
Statistical Analysis 3: Comparison: Flunisolide 320 mcg Per Day Pretreatment - Baseline vs Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.582, Mixed Models Analysis

3. Primary Outcome: Spirometry Forced Expiratory Flow 25-75% (FEF 25-75%)
Description: Indirectly assess small airway function.
Time Frame: baseline and six week followup
Population: Those subjects that completed the study protocol.
Measure: Mean (Standard Deviation); unit: % of predicted
Groups:
- Flunisolide 160 mcg Per Day Pretreatment - Baseline: Baseline in Patients who received inhaled Flunisolide HFA 80 mcg twice per day for a total of 160 mcg per day over the 6 week study period
- Flunisolide 320 mcg Per Day Pretreatment - Baseline: Baseline in patients who received inhaled Flunisolide HFA 160 mcg twice per day for a total of 320 mcg per day over the 6 week study period
- Flunisolide 160 mcg Per Day Posttreatment - 6 Wks: Six week followup in Patients who received inhaled Flunisolide HFA 80 mcg twice per day for a total of 160 mcg per day over the 6 week study period
- Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks: Six week followup in patients who received inhaled Flunisolide HFA 160 mcg twice per day for a total of 320 mcg per day over the 6 week study period
Arm/Group | Flunisolide 160 mcg Per Day Pretreatment - Baseline | Flunisolide 320 mcg Per Day Pretreatment - Baseline | Flunisolide 160 mcg Per Day Posttreatment - 6 Wks | Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks
Number analyzed (Participants) | 10 | 9 | 10 | 9
% of predicted | 60.3 (20.0) | 61.5 (13.7) | 57.7 (12.1) | 65.2 (18.9)
Statistical Analysis 1: Comparison: Flunisolide 160 mcg Per Day Pretreatment - Baseline vs Flunisolide 160 mcg Per Day Posttreatment - 6 Wks; Test type: Equivalence — The primary aim is to compare the average change in spirometric values (FEV1 and FEF25-75%) and AX from baseline to Week 6 from participants randomized flunisolide HFA 1 inhalation BID and to flunisolide HFA 2 inhalations BID; p = .782, Mixed Models Analysis; generalized linear mixed-effects models (GLMM) using the identity link function and normal distribution were used
Statistical Analysis 2: Comparison: Flunisolide 160 mcg Per Day Posttreatment - 6 Wks vs Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .906, Mixed Models Analysis; generalized linear mixed-effects models (GLMM) using the identity link function and normal distribution were used
Statistical Analysis 3: Comparison: Flunisolide 320 mcg Per Day Pretreatment - Baseline vs Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .102, Mixed Models Analysis; generalized linear mixed-effects models (GLMM) using the identity link function and normal distribution were used

4. Primary Outcome: Impulse Oscillometry (IOS) Resistance 5 (R5)
Description: Resistance of the respiratory system at 5 Hz is a measure of total airway resistance. Elevated value is indicative of respiratory dysfunction.
Time Frame: initial visit and six week followup
Population: Only data for subjects who completed study are presented.
Measure: Mean (Standard Deviation); unit: cmH2O(L/s)
Arm/Group | Flunisolide 160 mcg Per Day Pretreatment - Baseline | Flunisolide 320 mcg Per Day Pretreatment - Baseline | Flunisolide 160 mcg Per Day Posttreatment - 6 Wks | Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks
Number analyzed (Participants) | 10 | 9 | 10 | 9
cmH2O(L/s) | 6.5 (2.0) | 5.8 (2.3) | 7.0 (1.4) | 6.0 (1.8)
Statistical Analysis 1: Comparison: Flunisolide 160 mcg Per Day Pretreatment - Baseline vs Flunisolide 160 mcg Per Day Posttreatment - 6 Wks; Test type: Equivalence — To assess the impact of flunisolide on small airway parameters using spirometry and impulse oscillometry and determine whether there is a dose-related difference (320 mcg vs 160 mcg) with flunisolide HFA in pediatric patients who have evidence of small airway obstruction; p = .620, Mixed Models Analysis; generalized linear mixed-effects models (GLMM) using the identity link function and normal distribution were used
Statistical Analysis 2: Comparison: Flunisolide 160 mcg Per Day Posttreatment - 6 Wks vs Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = .543, Mixed Models Analysis; generalized linear mixed-effects models (GLMM) using the identity link function and normal distribution were used
Statistical Analysis 3: Comparison: Flunisolide 320 mcg Per Day Pretreatment - Baseline vs Flunisolide 320 mcg Per Day Posttreatment - 6 Weeks; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = .6, Mixed Models Analysis; generalized linear mixed-effects models (GLMM) using the identity link function and normal distribution were used

ADVERSE EVENTS:
Time Frame: up to 6 weeks
Arm/Group | Flunisolide 160 mcg Per Day | Flunisolide 320 mcg Per Day
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flunisolide 160 mcg Per Day (N=10) | Flunisolide 320 mcg Per Day (N=9)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The small numbers of subjects who qualified and completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-02-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT02404103/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-02-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT02404103/Prot_SAP_003.pdf